CLINICAL TRIAL: NCT03577314
Title: Dental Health in Recurrent Miscarriage
Brief Title: Is There an Interaction Between Recurrent Miscarriage and Dental Health
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gul Yildiz Telatar, Principal Investigator, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 40465587-179
Record Dates: First submitted 2018-06-21; First posted 2018-07-05 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Oral Health; Miscarriage
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- miscarriage: Patients were aged from 18 to 35 years, 50 females who have history of at least two unexplained recurrent miscarriage below 20th week of pregnancy
  Interventions: Other: miscarriage
- healthy: 50 systemically healthy females with at least two normal births and no poor obstetric history such as preeclampsia and premature birth
  Interventions: Other: miscarriage

INTERVENTIONS:
Other: miscarriage — (ORTHOPANTOMOGRAPH® OP300 PANORAMIC, Instrumentarium Dental, Tuusula, Finland,63 kVp, 0.8 mA, 0.5 s).
  Other Names: Intraoral and Radiographic Dental Examination

SUMMARY:
Oral infections can trigger the production of pro-inflammatory mediators that may be risk factors for miscarriage. The investigators investigated whether oral health care patterns that may promote or alleviate oral inflammation were associated with the history of miscarriage in Turkish women.

DETAILED DESCRIPTION:
Power analysis was performed with the G-Power software package to determine sample size.

To cover possible data loss, 10% of a group were added to each group. Medical and dental examination will be performed both of control and experimental groups. In dental examination decayed, missing, or filled teeth (DMFT) index will be used according to World Health Organization (WHO 1997) criteria. All teeth were visually using the International Caries Detection and Assessment System (ICDAS-II).

To analyze the correlation between oral health status and miscarriage linear regression test and for comparison of both the groups (case and control), two sample t test and chi square test were used.

ELIGIBILITY:
Inclusion Criteria:

* history of at least two unexplained recurrent miscarriage below 20th week of pregnancy
* systemically healthy females with at least two normal births
* no poor obstetric history such as preeclampsia and premature birth

Exclusion Criteria:

* history of thyroid disease, hyperprolactinemia, antiphospholipid syndrome, systemic lupus erythematosus, autoimmune diseases, thrombophilia, diabetes mellitus, uterine/cervical abnormalities, polycystic ovary syndrome, active liver disease, cardiovascular disease, premature ovarian failure, acute or chronic upper respiratory tract diseases, IVF pregnancy, multiple pregnancy, preeclampsia, arterial or venous embolism, infection,
* habit of smoking, alcohol, drug or caffeine,
* abnormal embryo karyotype,
* infection with hepatitis B or C, and HIV,
* chromosomal abnormalities,
* dental fluorosis,
* fluoride supplements,
* orthodontic appliances,
* body mass index ≥ 30 kg / m2
* age of the partner is found to be over 40

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients were aged from 18 to 35 years, 100 females
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-05-15 (Estimated)

PRIMARY OUTCOMES:
recurrent miscarriage | below 20th week of pregnancy
  If abortion material is obtainable, it will be genetically evaluated for chromosomal abnormalities. At least 8 weeks after termination of pregnancy, karyotype analysis of both couples and thrombophilia panel ( Factor V Leiden, prothrombin gene mutation G20210A, protein S/Protein C/antithrombin deficiency and MTHFR mutations) in the study group will be requested.

SECONDARY OUTCOMES:
Dental Examination | 1 Day
  All teeth were visually using the International Caries Detection and Assessment System (ICDAS-II). The chosen sites were recorded as:
  0 = sound;
  1. = first visible sign of noncavitated lesion seen only when the tooth is dried;
  2. = visible noncavitated lesion seen when wet and dry;
  3. = microcavitation in enamel;
  4. = noncavitated lesion extending into dentine seen as an undermining shadow;
  5. = small cavitated lesion with visible dentine: less than 50% of surface;
  6. = large cavitated lesions with visible dentine in more than 50% of the surface.
Periodontal Examination | 1 Day
  A single calibrated examiner measured probing depth-PD, 0: healthy
  1. bleeding
  2. calculus 3:3.5-5.5 mm
  4: over 5.5 mm
Clinical attachment level | 1 Day
  A single calibrated examiner measured clinical attachment level- CAL, 0: 0-3 mm 1:4-5 mm 2:6-8 mm 3:over 8mm 4: 9-11 mm 5: over 12 mm
Plaque Examination | 1 Day
  A single calibrated examiner measured plaque (Pl) 0:no plaque
  1. A film of plaque
  2. soft deposit s within the gingival pocket
  3. Abundance of soft matter within the gingival pocket
Gingival Examination | 1 Day
  A single calibrated examiner measured gingival indices (GI) 0= Normal gingiva;
  1. Mild inflammation
  2. Moderate inflammation
  3. Severe inflammation
Bleeding Examination | 1 Day
  A single calibrated examiner measured bleeding on probing (BOP) 0: no bleeding
  1: bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Gül Yıldız Telatar, Principal Investigator — Recep Tayyip Erdogan University Dentistry Faculty
Locations (2):
- Turkey (Türkiye) (2):
  - Recep Tayyip Erdogan University Dentistry Faculty, Rize
  - Recep Tayyip Erdogan University Faculty of Medicine, Rize

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available within 6 months of study finishing

REFERENCES:
- [Background] Heimonen A, Janket SJ, Meurman JH, Furuholm J, Ackerson LK, Kaaja R. Oral health care patterns and the history of miscarriage. Oral Dis. 2008 Nov;14(8):734-40. doi: 10.1111/j.1601-0825.2008.01460.x. PMID 19193203
- See also: Institute of Dentistry, Oulu University and Hospital, Oulu, Finland — http://www.ncbi.nlm.nih.gov/pubmed/?term=Oral+health+care+patterns+and+the+history+of+miscarriage